CLINICAL TRIAL: NCT02539745
Title: Associations of Vitamin D Deficiency and Vitamin D Receptor Polymorphisms With the Risk of Primary Open-angle Glaucoma
Status: Completed | Type: Observational
Sponsor: Lv Yingjuan (Other)
Responsible Party: Sponsor-Investigator, Lv Yingjuan, department of ophthamology, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Other Study IDs: tjykdxykyy1
Record Dates: First submitted 2015-08-03; First posted 2015-09-03 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Vitamin D Deficiency; Primary Open- Angle Glaucoma
Keywords: vitamin D; primary open- angle glaucoma
MeSH Terms: conditions — Vitamin D Deficiency; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cdx-2, Fok I, Bsm I and Taq I polymorphisms
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- primary open-angle glaucoma patients: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by enzyme-linked immunoabsorbent assay and vitamin D receptor polymorphic analysis was studied by real-time polymerase-chain reaction high resolution melting analysis in primary open-angle glaucoma patients.
  Interventions: Other: Vitamin D receptor polymorphic analysis; Other: Serum levels of 1a, 25-Dihydroxyvitamin D3
- randomly age-matched people: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by enzyme-linked immunoabsorbent assay and vitamin D receptor polymorphic analysis was studied by real-time polymerase-chain reaction high resolution melting analysis in randomly age-matched people.
  Interventions: Other: Vitamin D receptor polymorphic analysis; Other: Serum levels of 1a, 25-Dihydroxyvitamin D3

INTERVENTIONS:
Other: Vitamin D receptor polymorphic analysis — Vitamin D receptor polymorphic analysis was studied by real-time polymerase-chain reaction high resolution melting analysis.
Other: Serum levels of 1a, 25-Dihydroxyvitamin D3 — Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by enzyme-linked immunoabsorbent assay.

SUMMARY:
This study investigated whether vitamin D receptor gene polymorphism is altered in primary open-angle glaucoma subjects carrying the risk allele and vitamin D deficiency is an important factor in the development of glaucoma. Primary open-angle glaucoma patients and age-matched people in the Han population were enrolled. Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by enzyme-linked immunoabsorbent assay. Vitamin D receptor polymorphic analysis was studied by real-time polymerase-chain reaction high resolution melting analysis.

ELIGIBILITY:
Inclusion Criteria:

* intraocular pressure greater than 22 mmHg with two or more medications
* wide anterior chamber angle
* glaucomatous optic neuropathy (Glaucomatous optic nerve damage was defined as cup-to-disc ratio higher than 0.7 or focal loss of the nerve fiber layer (notch) associated with a consistent glaucomatous visual field defect)
* visual field loss consistent with optic nerve damage and visual fields were performed by using standard automated perimetry

Exclusion Criteria:

* the presence of any secondary glaucoma including exfoliation syndrome or a history of ocular trauma
* high myopia
* macular degeneration
* other ocular diseases
* a known history of systemic diseases and administration of vitamin D3 or other analog

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary open-angle glaucoma patients and randomly age-matched people as controls in the Han population of Tianjin China
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Serum levels of 1a, 25-Dihydroxyvitamin D3 | 1 day visit

SECONDARY OUTCOMES:
gene polymorphisms of vitamin D receptor | 1 day visit

CONTACTS AND LOCATIONS:
Overall Officials: xiaorong li, Study Director — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Lv Y, Yao Q, Ma W, Liu H, Ji J, Li X. Associations of vitamin D deficiency and vitamin D receptor (Cdx-2, Fok I, Bsm I and Taq I) polymorphisms with the risk of primary open-angle glaucoma. BMC Ophthalmol. 2016 Jul 19;16:116. doi: 10.1186/s12886-016-0289-y. PMID 27435453